CLINICAL TRIAL: NCT02596243
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Phase 2 Clinical Trial to Evaluate the Efficacy and the Safety of GX-188E, a DNA-based Therapeutic Vaccine, Administered Intramuscularly by Electroporation(EP) in HPV Type 16 and/or 18 Positive Patients With Biopsy-proven Cervical Intraepithelial Neoplasia Grade 2(CIN2), Grade 2/3 (CIN2/3), Grade 3(CIN3)
Brief Title: Phase 2 Clinical Trial to Evaluate the Safety and Efficacy of Plasmid DNA Therapeutic Vaccine(GX-188E)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HPV-EU-001
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: CIN2, CIN2/3, CIN3; Cervical Intraepithelial Neoplasia; High-Risk HPV; HPV infection; precancer Diseases; Double Blind; Safety/Efficacy
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections | interventions — GX-188 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GX-188E (Experimental): GX-188E + EP
  Interventions: Biological: GX-188E
- placebo (Placebo Comparator): Placebo + EP
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GX-188E — 1mg of GX-188E administered IM using EP device at day 0, week 4 and week 12.
  Other Names: DNA therapeutic vaccine
  Arms: GX-188E
Biological: Placebo — 0.5mL of Placebo administered IM using EP device at day 0, week 4 and week 12.
  Other Names: Placebo-control
  Arms: placebo

SUMMARY:
The purpose of this study is to access the efficacy and safety of GX-188E according the protocol in patients with Cervical Intraepithelial Neoplasia 2, 2/3 or 3 (CIN3)

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects age 18-60 years
2. Histologically confirmed HPV-16 or HPV-18 asspcoated CIN2, CIN 2/3 or CIN3 from tissue collected less than 10 weeks prior to Vaccination/EP #1 with overall lesion sizes less than 50% of the cervix area and no evidence of invasive cancer in any specimen;
3. Colposcopy is satisfactory based on visualization of the entire squamocolumnar junction and the upper limit of the entire aceto-white or suspected CIN disease area;
4. Healthy subjects as judged by the Investigator based on medical history, PE, and normal results for an ECG, CBC, Serum Chemistries, CPK and urinalysis done up to 4 weeks prior to enrolment;
5. For women who are not postmenopausal (at least 12 months of nontherapy- induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use a highly effective method of contraception during the treatment period and throughout Week 36 response evaluation visit.
6. Able and willing to comply with all study procedures and voluntarily signs informed consent form.

Exclusion Criteria:

1. Unsatisfactory colposcopy defined as incomplete visualization of the entire squamocolumnar junction and the upper limit of the entire aceto-white or suspected CIN disease area;
2. Pregnancy or breastfeeding;
3. Immunosuppression including any concurrent condition requiring the continued use of systemic or topical steroids at or near the injection site [deltoid, upper arm] (excluding inhaled and eye drop-containing corticosteroids) or the use of immunosuppressive agents. All other corticosteroids must be discontinued > 4 weeks prior to Day 0 of study vaccine administration; autoimmune disorders, transplant recipients;
4. History of previous therapeutic HPV vaccination (individuals who have been immunized with licensed prophylactic HPV vaccines (e.g. Gardasil®, Cervarix®) are not excluded);
5. Positive serological test for hepatitis C virus or hepatitis B virus surface antigen (HBsAg) or human immunodeficiency virus (HIV);
6. Administration of any blood product within 3 months of enrollment;
7. Administration of any licensed vaccine within 2 weeks of enrollment (4 weeks for measles vaccine);
8. Participation in a study with an investigational compound or device within 30 days prior to signing informed consent;
9. Cardiac pre-excitation syndromes (such as Wolff-Parkinson-White);
10. History of seizures (unless seizure free for 5 years);
11. Tattoos, scars, active lesions/rashes or any implantable leads within 3 cm of the intended site of vaccination/EP;
12. Any electronic medical implants (such as cardiac pacemaker);
13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements;
14. A tendency for severe haemorrhage following acute trauma;
15. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (i.e. infections disease) illness must not be enrolled into this study;
16. Any other conditions judged by the investigator that would limit the evaluation of a subject.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with histopathological regression of cervical lesions to CIN1 or less | 36 weeks
  The number of participants with cervical lesions regress to CIN1 or less at the 36 week visit

SECONDARY OUTCOMES:
Number of participants with Clearance of HPV 16 or 18 in combination with histopathological regression of cervical lesions to CIN1 or less | 36 weeks
  The number of participants with clearance of HPV 16 or 18 in combination with histopathological regression of cervical lesions to CIN1 or less at the 36 week visit

CONTACTS AND LOCATIONS:
Overall Officials: Terje Raud, MD, Principal Investigator — Tartu University Hospital; Kersti Kukk, MD, Principal Investigator — North Estonia Medical Centre Foundation; Aira Peri, MD, Principal Investigator — East Tallinn Central Hospital; Tetiana Tatarchuk, MD, Principal Investigator — National Academy of Medical Sciences of Ukraine; Nataliya Lutsenko, MD, Principal Investigator — State Institution, Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine; Sergiy Kartashov, MD, Principal Investigator — Kharkiv medical academy of postgraduate education; Natalia Rozhkovska, MD, Principal Investigator — Multi-profile Medical Center (University Clinic No. 1) of Odesa National Medical University
Locations (16):
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- South Korea (9):
  - Inje University Busan Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Severance Hospital, Seoul
  - Cheil General Hospital & Women's Healthcare Center, Seoul
  - CHA Gangnam Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ehwa Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Ukraine (4):
  - Kharkiv medical academy of postgraduate education, Kharkiv
  - National Academy of Medical Sciences of Ukraine, Kyiv
  - Multi-profile Medical Center (University Clinic No. 1) of Odesa National, Odesa
  - State Institution Zaporizhzhia Medical Academy of Post-Graduate Education, Zaporizhzhya